CLINICAL TRIAL: NCT06890793
Title: Comparative Analysis of Heart Rate Variability in Patients with Cervical Pain, Lumbar Pain, and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Clinical Professor, Universidad de Extremadura
Other Study IDs: 09
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low Back Pain (CLBP); Chronic Neck Pain; Heart Rate Variability; Autonomic Nervous System Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Subjects: This group includes adults aged 18-65 years without any chronic or acute pathology, no regular medication that could alter autonomic nervous system function, and no low back pain in the past six months.
- Chronic Low Back Pain Subjects: This group includes adults aged 18-65 years diagnosed with chronic low back pain lasting at least three months, with a minimum pain intensity of 3/10 on the Numerical Pain Rating Scale, and without uncontrolled neurological or cardiac disorders.
- Chronic Neck Pain Subjects: This group includes adults aged 18-65 years diagnosed with chronic neck pain lasting at least three months, with a minimum pain intensity of 3/10 on the Numerical Pain Rating Scale, and without uncontrolled neurological or cardiac disorders.

SUMMARY:
This is a cross-sectional study designed to evaluate potential differences in heart rate variability (HRV) indices based on the affected body region (cervical vs lumbar) in individuals with chronic pain. The study will compare HRV parameters between three groups: individuals with chronic neck pain (CNP), individuals with chronic low back pain (CLBP), and a control group without pain. HRV will be assessed using a Firstbeat Bodyguard® device over a 10-minute period, and the data will be analyzed with Kubios® HRV software. The study aims to determine whether autonomic nervous system modulation differs depending on the location of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* - Adults aged between 18 and 65 years.

For the chronic low back pain group:

* Diagnosis of chronic neck or low back pain lasting at least three months.
* A minimum pain intensity of 3/10 on the Numerical Pain Rating Scale (NPRS).

For the healthy group:

* Absence of any chronic or acute pathology.
* No regular medication that could alter autonomic nervous system function.
* No episodes of low back pain in the past six months.

Exclusion Criteria:

* Presence of uncontrolled neurological or cardiac disorders.
* Use of medications that could influence autonomic function or pain perception (e.g., opioids, antidepressants, benzodiazepines, anti-inflammatory drugs, beta-blockers) within two weeks prior to the study.
* Body Mass Index (BMI) equal to or greater than 30 kg/m².

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include three groups: one group of adults diagnosed with chronic neck pain (CNP), one group of adults diagnosed with chronic low back pain (CLBP), and another group of healthy adults within the same age range. Participants will be recruited from local community advertisements and hospital outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Root Mean Square of Successive Differences (rMSSD) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  This variable represents a time-domain measure of heart rate variability, reflecting parasympathetic nervous system activity and short-term variability in R-R intervals. It is calculated as the root mean square of differences between successive R-R intervals. rMSSD is an established metric to assess vagal modulation and is sensitive to changes in autonomic function.
Standard Deviation 1 (SD1) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  A non-linear metric derived from the Poincaré plot of heart rate variability, indicating short-term variability in R-R intervals. It is closely associated with parasympathetic activity and vagal modulation.
Standard Deviation 2 (SD2) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  A non-linear metric derived from the Poincaré plot, representing long-term variability in R-R intervals. SD2 is inversely related to sympathetic activity and reflects the balance between sympathetic and parasympathetic modulation.
Stress Score (SS) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  This variable is calculated as the reciprocal of SD2, multiplied by 1000. It reflects the level of sympathetic activation, where higher Stress Score values indicate increased stress and reduced parasympathetic activity.
Sympathetic/Parasympathetic Ratio (S/PS Ratio) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  This variable represents the ratio of Stress Score to SD1. It reflects the balance between sympathetic and parasympathetic modulation, with higher values indicating sympathetic dominance, commonly observed in chronic pain conditions.

SECONDARY OUTCOMES:
Mean Heart Rate (Mean HR) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  Represents the average heart rate (beats per minute) recorded during the data collection period. It serves as a general indicator of autonomic activity, providing insights into the balance between sympathetic and parasympathetic modulation.
Minimum Heart Rate (Min HR) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  Represents the lowest heart rate (beats per minute) recorded during the data collection period. This variable reflects periods of parasympathetic predominance and is useful for assessing vagal.
Maximum Heart Rate (Max HR) | Measured during a single 30-minute session, including a 5-minute baseline and 25-minute data collection period.
  Represents the highest heart rate (beats per minute) recorded during the data collection period. This variable reflects periods of sympathetic activation and provides insights into stress responses during the session.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antúnez, Ph.D., Study Director — University of Extremadura
Locations (1):
- Universidad de Extremadura, Badajoz, Badajoz, Spain